CLINICAL TRIAL: NCT04781010
Title: Characterization and Outcome of Children With Leukodystrophy: An Observational Study at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagat Mohamed Shehata, assistant specialist, Sohag University
Other Study IDs: Soh-Med-21-02-01
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Children With Leukodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — MRI pattern in children with Leukodystrophy

SUMMARY:
Leukodystrophies are heterogeneous genetic disorders characterized by the selective involvement of white matter in the central nervous system (CNS) (1, 2). Inherited leukodystrophies are diseases of the myelin, including abnormal myelin development, hypomyelination, or degeneration of myelin (3, 4).

Most of these disorders fall into one of three categories; lysosomal storage diseases, peroxisomal disorders, and diseases caused by mitochondrial dysfunction and each leukodystrophy has distinctive clinical, biochemical, pathologic, and radiologic features (5).

ELIGIBILITY:
Inclusion Criteria:

* The patients fulfilling all the following criteria will be included:

  1. Age ≤ 18 years.
  2. The presence of typical clinical, biochemical, and neuroimaging features of leukodystrophies.

Exclusion Criteria:

* 1- Children who have coexistent genetic disorders. 2- Children who have cerebral malformations. 3- History of perinatal asphyxia. 4- History of head trauma or intracranial hemorrhage. 5- Acquired CNS myelin disorders, such as multiple sclerosis and related acquired demyelinating processes, infectious and post-infectious white matter damage, toxic injuries and non-genetic vascular insults.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include children with leukodystrophy diagnosed and followed-up at the pediatric neurology clinic of Sohag University Hospital during the period of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
White matter changes in MRI | 2 years
  Brain MRI of all patients will be systematically reviewed, particularly Sagittal T1, Axial T1, T2-weighted and fluid-attenuated inversion-recovery (FLAIR) sequences. Other sequences will be also reviewed if available, such as MR spectroscopy (MRS) (for mitochondrial disorders or Canavan disease to investigate abnormalities in lactate or N-acetyl aspartate (NAA) respectively), and diffusion-weighting (useful in disorders such as AARS2-related leukoencephalopathy).
Biochemical changes | 2 years
  1. Arylsulfatase A levels can be measured in the leukocytes if suspected Metachromatic Leukodystrophy.
  2. Galactocerebrosidase (GALC) enzyme level for Krabbe's Disease.
  3. Plasma VLCFAs for Adrenoleukodystrophy.
  4. NAA levels in the urine for Canavan's Disease.
  5. Beta galactosidase in leukocytes deficient in cases of infantile GM1 gangliosidosis &Hexosaminidase for Tay Sachs disease.
  6. Plasma FSH ,LH markedly reduced in cases of 4 H (Hypomyelination, hypodontia and hypogonadotropic hypogonadism syndrome).
  7. Genetic testing for certain diseases

SECONDARY OUTCOMES:
Electrophysiological changes | 2 years
  including nerve conduction studies and electromyography will be useful in identifying peripheral nerve involvement (e.g., in AMN, MLD, Krabbe) or myopathy with or without a neuropathy (e.g., in mitochondrial diseases) or metachromatic leukodystrophy. Moreover, electroencephalographic data will be assessed, particularly in patients with seizures.
Tandem mass spectrometry (MS/MS) finding | 2 years
  We will obtain patients' blood samples on a Glutheric card, Acylcarnitines and amino acids will be analysed using ACQUTIY TQD Tandem quadrupole UPLC/MS/MS with apositive electrospray ionization prope according to the manufacturer's instructions.
Urinary organic acid analysis | 2 years
  by GC/MS using agilent 7890 and 5975 systems. Results will be calculated in mol/mmol creatinine using acalipration curve of the organic acid of interest that will be processed under the same conditions.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Parikh S, Bernard G, Leventer RJ, van der Knaap MS, van Hove J, Pizzino A, McNeill NH, Helman G, Simons C, Schmidt JL, Rizzo WB, Patterson MC, Taft RJ, Vanderver A; GLIA Consortium. A clinical approach to the diagnosis of patients with leukodystrophies and genetic leukoencephelopathies. Mol Genet Metab. 2015 Apr;114(4):501-515. doi: 10.1016/j.ymgme.2014.12.434. Epub 2014 Dec 29. PMID 25655951
- [Result] Berger J, Moser HW, Forss-Petter S. Leukodystrophies: recent developments in genetics, molecular biology, pathogenesis and treatment. Curr Opin Neurol. 2001 Jun;14(3):305-12. doi: 10.1097/00019052-200106000-00007. PMID 11371752